CLINICAL TRIAL: NCT06063239
Title: Probiotics in Special Needs Patients at High Risk for Tooth Decay: a Randomized Controlled Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Prof. Marco Dolci, MD DDS PHD, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CARIES
Record Dates: First submitted 2023-09-26; First posted 2023-10-02 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Tooth Decay; Intellectual Disability; Caries,Dental
Keywords: caries;; tooth decay; intellectual disability; probiotics; lactobacillus rhamnosus; lactobacillus plantarum; pH
MeSH Terms: conditions — Dental Caries; Intellectual Disability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: SNOSE Sequentially Numbered, Opaque, Sealed Envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Group (Experimental): Subjects who will receive orally administred probiotics based on L. rhamnosus and L. plantarum for 90 days in adjunction to the instruction of their care-giver regarding oral hygiene procedures.
  Interventions: Other: Test Group
- Positive Control (Active Comparator): Subjects who will receive orally administred probiotics based on placebo for 90 days in adjunction to the instruction of their care-giver regarding oral hygiene procedures.
  Interventions: Other: Positive Control
- Negative Control (Other): Subjects who will receive esclusively the instruction of their care-giver regarding oral hygiene procedures.
  Interventions: Other: Negative Control

INTERVENTIONS:
Other: Test Group — Subjects will receive orally administred probiotics based on L. plantarum and L. rhamnosus for 90 days
  Arms: Test Group
Other: Positive Control — Subjects will receive orally administred probiotics based on placebo 90 days
  Arms: Positive Control
Other: Negative Control — Subjects will receive esclusively instruction to perform oral hygiene procedures properly.
  Arms: Negative Control

SUMMARY:
The goal of this randomized clinical trial is to test the effect orally administration of Probiotics based on Lactobacillus rhamnosus LR04 and Lactobacillus plantarum LP14 as adjuvant in caries prevention in subjects who can not properly perform oral hygiene procedures. The main questions it aims to answer are:

* QUESTION 1: orally administered probiotics based on the previous strains could represent a useful tool in support of special needs patients in tooth decay prevention?
* QUESTION 2: orally administered probiotics based on the previous strains could ameliorate salivary pH management?

Partecipants in the test group will take the test probiotic for 90 days in adjunction of the routinary oral hygiene procedures.

Partecipants in the positive controlled group will take the placebo for 90 days in adjunction of the routinary oral hygiene procedures.

Partecipants in the negative control group will perform only the routinary oral hygiene procedures.

Researchers will compare 3 groups to see if orally administered probiotics based on L. rhamnosus and L. plantarum may help in the management of clinical status and salivary pH levels.

DETAILED DESCRIPTION:
Recent literature has highlighted how patients' oral health is closely linked to the presence of intellectual and developmental disabilities (IDD). It has in fact been found that in patients with IDD the level of oral health tends to be lower than in subjects without IDD, and how this has an influence on the general state of health. A key role appears to be played by caregivers, who carry out the delicate task of maintaining an adequate level of oral hygiene. Among various aspects, daily oral hygiene maneuvers were considered as a key intervention in maintaining good health. In this regard, it is worth remembering that a study conducted in 1990 on caregivers demonstrated how, despite knowing the characteristics of the healthy appearance of the tissues supporting the dental elements, not everyone knew how this was closely related to the oral hygiene. Likewise, the study by Kilian and collaborators demonstrated how the maintenance of an oral microbiota that promotes oral health is not only desirable, but also possible. Given that the implementation of correct home hygiene represents a cornerstone in the management of general well-being, we decided to evaluate whether a formulation that allows the strengthening of bacterial populations competitive with respect to cariogenic populations could be significantly useful for the maintenance of these patients.

Inclusion criteria: adult and minor special needs patients belonging to the University Dental Clinic of Chieti. Presence of motor and/or cognitive difficulties in carrying out oral hygiene maneuvers at home.

Exclusion criteria: special needs patients with effective home hygiene.

Minimum sample size: Calculation of sample size (Alpha = 0.05; Power = 95%) for 3 independent study groups, and a continuous primary endpoint.

Sample size = Z2 (1-alpha/2) p (1-p) / d2 Where Z(1-alpha/2) is the standard variate corresponding to 1.96 at 5% type 1 error, p is the expected proportion in the population expressed in decimals based on previous studies and d is the confidence level decided by the researcher expressed in decimal. 20 patients are required per group, for a total of 60 patients. To these patients, the dropout percentage of 10% must be added, so the total is 70 patients.

BASELINE - T0. Signature of informed consent. Completion of a specific questionnaire regarding consumption of simple sugars and initial home oral hygiene procedures. Oral cavity inspection with registration of gingivitis according to dichotomous qualitative indices by quadrants.Recording of specific parameters: Salivary pH via GEASS® pH meter. DMFT (Decayed Missing Filled Teeth).

Random placement of the patient in the test, positive or negative control group.

TEST: instruction of the subject and/or caregiver in home oral hygiene 2/day + oeally administred probiotic based on L. plantarum and L. rhamnosus for 90 days.

POSITIVE CONTROL: instruction of the subject and/or caregiver in home oral hygiene 2/day + orally administred placebo.

NEGATIVE CONTROL: instruction of the subject and/or caregiver for home oral hygiene procedures 2/day.

T1 - AFTER 3 MONTHS FROM T0. Oral cavity inspection with recording of gingivitis according to dichotomous qualitative indices by quadrants. Recording of pH and DMFT.

Randomization. The treatment that is due to the individual patient is kept in sequentially numbered, opaque and sealed envelopes (SNOSE Sequentially Numbered, Opaque, Sealed Envelopes). The products used for both the test and the controls will be supplied in anonymous tubes so that neither the patient nor the investigator will be aware of them.

Statistical analysis: Developed by trusted bioinformatics group.

ELIGIBILITY:
Inclusion Criteria:

* individuals with intellectual disability in presence of gingivitis in 1 quadrant at least and 1 decayed tooth at least, and improper oral hygiene routine.

Exclusion Criteria:

* individuals without intellectual disability or with the condition in absence of gingivitis, decayed teeth and improper oral hygiene routine.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of clinical dicotomic indexes for gingivitis | From enrollement to the end of treatment at 3 months.
  Gingivitis will be recorded for each quadrant as present/absent taking into account the classical flogistic signs.

SECONDARY OUTCOMES:
management of salivary pH | From enrollement to the end of treatment at 3 months.
  Salivary pH will be recorded via digital pHmeter 3/times for each time-point in order to minimaze the error of registration.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Dolci, MD DDS PHD, Principal Investigator — University G. d'Annunzio of Chieti
Locations (1):
- University G. d'Annunzio, Chieti, Italy

IPD SHARING:
Plan to Share IPD: No
A decision regarding IPD sharing has not been made yet because a dedicated website is not available at the momente.

REFERENCES:
- [Background] Wilson NJ, Lin Z, Villarosa A, Lewis P, Philip P, Sumar B, George A. Countering the poor oral health of people with intellectual and developmental disability: a scoping literature review. BMC Public Health. 2019 Nov 15;19(1):1530. doi: 10.1186/s12889-019-7863-1. PMID 31729967
- [Background] Mac Giolla Phadraig C, Farag M, McCallion P, Waldron C, McCarron M. The complexity of tooth brushing among older adults with intellectual disabilities: Findings from a nationally representative survey. Disabil Health J. 2020 Oct;13(4):100935. doi: 10.1016/j.dhjo.2020.100935. Epub 2020 May 11. PMID 32439304
- [Background] Minihan PM, Morgan JP, Park A, Yantsides KE, Nobles CJ, Finkelman MD, Stark PC, Must A. At-home oral care for adults with developmental disabilities: a survey of caregivers. J Am Dent Assoc. 2014 Oct;145(10):1018-25. doi: 10.14219/jada.2014.64. PMID 25270700
- [Background] Waldron C, Nunn J, Mac Giolla Phadraig C, Comiskey C, Guerin S, van Harten MT, Donnelly-Swift E, Clarke MJ. Oral hygiene interventions for people with intellectual disabilities. Cochrane Database Syst Rev. 2019 May 31;5(5):CD012628. doi: 10.1002/14651858.CD012628.pub2. PMID 31149734
- [Background] Molina G, Zar M, Dougall A, McGrath C. Management of dental caries lesions in patients with disabilities: Update of a systematic review. Front Oral Health. 2022 Oct 28;3:980048. doi: 10.3389/froh.2022.980048. eCollection 2022. PMID 36389277
- [Background] Petrovic BB, Peric TO, Markovic DLJ, Bajkin BB, Petrovic D, Blagojevic DB, Vujkov S. Unmet oral health needs among persons with intellectual disability. Res Dev Disabil. 2016 Dec;59:370-377. doi: 10.1016/j.ridd.2016.09.020. Epub 2016 Sep 30. PMID 27697655
- [Background] Al-Maweri SA, Zimmer S. Oral Health Survey of 6-14-Year-Old Children with Disabilities Attending Special Schools Yemen. J Clin Pediatr Dent. 2015 Spring;39(3):272-6. doi: 10.17796/1053-4628-39.3.272. PMID 26208074
- [Background] Nqcobo CB, Yengopal V, Rudolph MJ, Thekiso M, Joosab Z. Dental caries prevalence in children attending special needs schools in Johannesburg, Gauteng Province, South Africa. SADJ. 2012 Aug;67(7):308-13. PMID 23951782
- [Background] Uwayezu D, Gatarayiha A, Nzayirambaho M. Prevalence of dental caries and associated risk factors in children living with disabilities in Rwanda: a cross-sectional study. Pan Afr Med J. 2020 Jul 17;36:193. doi: 10.11604/pamj.2020.36.193.24166. eCollection 2020. PMID 32952837
- [Background] Jang HJ, Kim JH, Lee NK, Paik HD. Probiotic Lactobacillus plantarum Ln4 Showing Antimicrobial and Antibiofilm Effect against Streptococcus mutans KCTC 5124 Causing Dental Caries. J Microbiol Biotechnol. 2024 Jan 28;34(1):116-122. doi: 10.4014/jmb.2306.06001. Epub 2023 Sep 8. PMID 37674399
- [Background] Butt S, Sin M. Can probiotics prevent dental caries? Evid Based Dent. 2023 Sep;24(3):130-131. doi: 10.1038/s41432-023-00918-z. Epub 2023 Sep 5. PMID 37670134
- [Background] Teanpaisan R, Surachat K, Wonglapsuwan M, Piwat S, Pahumunto N. Short-term use of Lacticaseibacillus rhamnosus SD11 and the oral microbiome: Low caries RCT study. Oral Dis. 2024 May;30(4):2736-2745. doi: 10.1111/odi.14681. Epub 2023 Jul 16. PMID 37455386
- [Background] Porksen CJ, Keller MK, Damholt A, Frederiksen AKS, Ekstrand KR, Markvart M, Larsen T, Bakhshandeh A. The effect of a lozenge combining prebiotic arginine and probiotics on caries increment in children during 10-12 months, a randomized clinical trial. J Dent. 2023 Aug;135:104599. doi: 10.1016/j.jdent.2023.104599. Epub 2023 Jun 24. PMID 37356561
- [Background] Meng N, Liu Q, Dong Q, Gu J, Yang Y. Effects of probiotics on preventing caries in preschool children: a systematic review and meta-analysis. J Clin Pediatr Dent. 2023 Mar;47(2):85-100. doi: 10.22514/jocpd.2023.014. Epub 2023 Mar 3. PMID 36890746
- [Background] Zeng Y, Fadaak A, Alomeir N, Wu TT, Rustchenko E, Qing S, Bao J, Gilbert C, Xiao J. Lactobacillus plantarum Disrupts S. mutans-C. albicans Cross-Kingdom Biofilms. Front Cell Infect Microbiol. 2022 Mar 22;12:872012. doi: 10.3389/fcimb.2022.872012. eCollection 2022. PMID 35392605
- [Background] Jung HY, Cai JN, Yoo SC, Kim SH, Jeon JG, Kim D. Collagen Peptide in a Combinatorial Treatment with Lactobacillus rhamnosus Inhibits the Cariogenic Properties of Streptococcus mutans: An In Vitro Study. Int J Mol Sci. 2022 Feb 7;23(3):1860. doi: 10.3390/ijms23031860. PMID 35163782
- [Background] Gonczi NN, Strang O, Bagi Z, Rakhely G, Kovacs KL. Interactions between probiotic and oral pathogenic strains. Biol Futur. 2021 Dec;72(4):461-471. doi: 10.1007/s42977-021-00091-3. Epub 2021 Jun 2. PMID 34554489
- [Background] Pahumunto N, Piwat S, Chanvitan S, Ongwande W, Uraipan S, Teanpaisan R. Fermented milk containing a potential probiotic Lactobacillus rhamnosus SD11 with maltitol reduces Streptococcus mutans: A double-blind, randomized, controlled study. J Dent Sci. 2020 Dec;15(4):403-410. doi: 10.1016/j.jds.2020.03.003. Epub 2020 May 6. PMID 33505609
- [Background] Tahmourespour A, Kasra-Kermanshahi R, Salehi R. Lactobacillus rhamnosus biosurfactant inhibits biofilm formation and gene expression of caries-inducing Streptococcus mutans. Dent Res J (Isfahan). 2019 Mar-Apr;16(2):87-94. PMID 30820202